CLINICAL TRIAL: NCT04722523
Title: A Pilot Study of Neoadjuvant Cemiplimab With Platinum-Doublet Chemotherapy, and Cetuximab in Patients With Resectable, Locally Advanced Head and Neck Squamous Cell Carcinoma
Brief Title: A Study of Cemiplimab With Chemotherapy and Immunotherapy in People With Head and Neck Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 20-445
Record Dates: First submitted 2021-01-21; First posted 2021-01-25 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Head and Neck Cancer; Head Cancer; Head Cancer Neck; Neck Cancer; Head and Neck Squamous Cell Carcinoma; HNSCC
Keywords: Cemiplimab; Platinum-Doublet Chemotherapy; Cetuximab; Head and Neck Cancer; Head Cancer; Neck Cancer; Head and Neck Squamous Cell Carcinoma; Memorial Sloan Kettering Cancer Center; 20-445; HNSCC)
MeSH Terms: conditions — Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck | interventions — Cisplatin; Carboplatin; Docetaxel; Cetuximab; cemiplimab; Paclitaxel

STUDY DESIGN:
Intervention Model Description: Six patients can be enrolled once the study has opened to the starting dose level. If 0-1 of the first 6 patients treated on study experience a DLT, then an additional 4 patients will be accrued to the study. If 0-2 of the 10 patients experience a DLT, then the combination will be deemed to be safe. If >2 of the first 6 patients accrued or >3 of 10 patients accrued experience a DLT, then patients will be treated at one dose level reduction.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Head and Neck Squamous Cell Cancer/HNSCC (Experimental): Participants with locally advanced, resectable head and neck squamous cell carcinoma for which standard-of-care management would entail definitive surgery followed by adjuvant radiation +/- concurrent chemotherapy are eligible.
  Interventions: Drug: Cisplatin; Drug: Carboplatin; Drug: Docetaxel; Drug: Cetuximab; Drug: Cemiplimab; Procedure: Surgical Resection of Primary +/- Neck Dissection; Radiation: Post-operative radiation therapy; Drug: Paclitaxel
- Secondary Cohort (Experimental): Participants with locally advanced, resectable head and neck squamous cell carcinoma for which standard-of-care management would entail definitive surgery followed by adjuvant radiation +/- concurrent chemotherapy are eligible.
  Interventions: Drug: Cetuximab; Drug: Cemiplimab

INTERVENTIONS:
Drug: Cisplatin — Cisplatin 75mg/m2 AUC 5 on weeks 2, 5, and 8
  Arms: Head and Neck Squamous Cell Cancer/HNSCC
Drug: Carboplatin — Carboplatin AUC 5 on weeks 2, 5, and 8
  Arms: Head and Neck Squamous Cell Cancer/HNSCC
Drug: Docetaxel — Docetaxel 75mg/m2 on weeks 2, 5, and 8
  Arms: Head and Neck Squamous Cell Cancer/HNSCC
Drug: Cetuximab — Cetuximab 400mg/m2 on week 1, 250mg/m2 on weeks 2, 3, 4, 5, 6, 7, 8, 9, 10
Drug: Cemiplimab — Cemiplimab 350mg on weeks 2, 5, 8, 11; if adjuvant radiation +/- chemotherapy is omitted, Cemiplimab will be administered on weeks 16, 19, 22, 25, 28, 31, 34, 37
Procedure: Surgical Resection of Primary +/- Neck Dissection — Twenty-eight days (+ 7 days) following the 3rd cycle of neoadjuvant therapy, patients will then undergo definitive surgical resection of the primary site +/- neck dissection(s).
  Arms: Head and Neck Squamous Cell Cancer/HNSCC
Radiation: Post-operative radiation therapy — Post-operative radiation therapy +/- radiosensitizing agent(s) will be administered per standard-of-care based on pathologic staging of the surgical specimen. If there is an excellent response to treatment with a high degree of downstaging the addition of adjuvant radiation may be omitted if NCCN guidelines are met. If the pathologic stage following induction systemic therapy and surgery is ypT1-2N0 without the presence of adverse features that include positive margins or a combination of perineural invasion, vascular invasion, and a depth of invasion of >0.5mm, adjuvant radiation will not be administered, consistent with the NCCN guidelines [2]. Otherwise, patients will receive adjuvant RT-based treatment with standard radiation techniques.
  Arms: Head and Neck Squamous Cell Cancer/HNSCC
Drug: Paclitaxel — If participants are unable to receive Docetaxel due to lack of insurance approval or due to an allergic reaction, Docetaxel can be substituted with Paclitaxel. Paclitaxel would be dosed at 90 mg/m2 on weeks 2, 3, 5, 6, 8 and 9.
  Other Names: Taxol
  Arms: Head and Neck Squamous Cell Cancer/HNSCC

SUMMARY:
The purpose of this study is to find out whether combining the standard chemotherapy for head and neck cancer with the immunotherapy drugs cetuximab and cemiplimab (the study drug) is a safe treatment for head and neck cancer, and whether receiving this combination treatment before surgery may allow participants to forgo the standard radiation treatment after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically (histologically or cytologically) proven diagnosis of squamous cell carcinoma of the head and neck that has arisen from the oral cavity, oropharynx, nasal cavity, paranasal sinuses, larynx, or hypopharynx
* Clinical stage T1, N2-3; T2, N1-3, T3/T4a, Any N (AJCC, 8th ed.) without evidence of distant metastasis (M0) based on PET/CT or CT chest, abdomen, and pelvis, for which standard-of-care treatment would entail surgical resection with adjuvant radiation +/- chemotherapy.

  ° Patients with recurrent and multiple primary head and neck cancers that are surgically resectable are eligible if the patient did not receive prior radiation or systemic therapy.
* Disease must be amenable to surgical resection.
* The patient must be a surgical candidate.

  1. Hemoglobin > 9.0 g/dL
  2. Absolute neutrophil count (ANC) >1.5 x 10^9/L
  3. Platelet count >100 x 10^9/L
  4. Serum creatinine <1.5 upper limit of normal (ULN) or estimated creatinine clearance (CrCl) >30 mL/min
  5. Adequate hepatic function:
* Total bilirubin <1.5 x upper limit of normal ULN)
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) both < 3 x ULN
* Alkaline phosphatase (ALP) <2.5 x ULN Note: For patients with Gilbert syndrome, total bilirubin <3x ULN. Upper central must be documented appropriately as past medical history.
* Men and woman >18 years old
* Eastern cooperative oncology group performance status < 1

Exclusion Criteria:

* Prior radiation and systemic therapy for a head and neck cancer.
* Oral cavity cancer that is not amenable to surgical resection or the patient is not a surgical candidate.
* Active or prior documented autoimmune or inflammatory disorders that have been treated with steroids or immunomodulator therapy in the past 5 years.

Exceptions: Patients with vitiligo, type 1 diabetes mellitus, and endocrinopathies (including hypothyroidism due to autoimmune thyroiditis) only requiring hormone replacement, childhood asthma that is resolved, or psoriasis it does not require systemic treatment are permitted.

* Conditions requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalents) or other immunosuppressant medications within 14 days of treatment on study.
* Receipt of live attenuated vaccine within 30 days prior initiating treatment on study.
* Prior allogeneic stem cell transplantation, or autologous stem cell transplantation.
* Any infection requiring hospitalization and/or intravenous antibiotic therapy within 2 weeks of the start of treatment.
* Uncontrolled infection with human immunodeficiency virus (HIV), hepatitis B or hepatitis C virus (HBV or HCV) infection; or diagnosis of immunodeficiency.

  1. Patients with known HIV infection who have controlled infection (undetectable viral load (HIV RNA PCR) and CD4 count above 350, either spontaneously or on a stable antiviral regimen) are permitted. For patients with controlled HIV infection monitoring will be performed per local standards
  2. Patients with HBV (hepatitis B surface antigen positive; HBsAg+) who have controlled infection (serum HBV DNA PCR that is below the limit of detection and receiving anti-viral therapy for HBV) are permitted. Patients with controlled infections must undergo periodic monitoring of HBV DNA. Patients must remain on anti-viral therapy for at least 6 months be on the last dose of Cemiplimab.
  3. Patients were HCV antibody positive (HCV Ab+) who have controlled infection (undetectable HCV RNA by PCR, either spontaneously or in response to successful prior course of anti-HCV therapy) are permitted.
* History of immune-related pneumonitis with the last 5 years.
* History of interstitial lung disease (e.g., idiopathic pulmonary fibrosis, organizing pneumonia) or active, noninfectious pneumonitis that required immune-suppressive doses of leuko-corticoids to assist with management.
* Known hypersensitivity or allergy to any of the excipients in the cemiplimab drug product.
* Patients with a history of solid organ transplant (exception: corneal transplant)
* Any medical comorbidity, physical examination finding, or metabolic dysfunction, or clinical laboratory abnormality that in the opinion of the investigator renders the patient unsuitable for participation in a clinical trial due to high safety risks.
* Women with a positive serum or urine beta-hCG pregnancy test at screening/baseline visit. If positive, pregnancy must be ruled out by ultrasound for patient to be eligible.
* Breast-feeding women
* Women of childbearing potential who are sexually active and aren't willing to practice highly effective contraception prior to the first dose of Cemiplimab, during the study, and for at least 180 days after the last dose. Highly effective contraceptive measures include:

  1. Stable use of combined estrogen and progesterone containing hormonal contraception or progesterone and-only hormonal contraception associated with inhibition of ovulation initiated 2 or more menstrual cycles prior to screening
  2. Intrauterine device; intrauterine hormone-releasing system
  3. Bilateral tubal ligation
  4. Vasectomized partner and/or
  5. Sexual abstinence

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-01-20 (Actual); Primary Completion 2026-06-20 (Estimated); Study Completion 2026-06-20 (Estimated)

PRIMARY OUTCOMES:
Incidence of toxicities graded according to NCI CTCAE | 1 year
  The primary endpoint is safety and tolerability, which will be evaluated by a description of observed adverse events by grades. All toxicities will be graded according to NCI CTCAE, Version5.0. The regimen will be deemed safe and well tolerated if there are 2 or fewer DLTs out of 10 patients enrolled. A DLT is defined as any non-hematologic grade 3 or greater adverse event as defined by CTCAE v5.0 that is thought to be related to the addition of Cemiplimab to the combination of a platinum-doublet with cetuximab.

CONTACTS AND LOCATIONS:
Overall Officials: Lara Dunn, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering Basking Ridge (Limited Protocol Activities), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (Limited Protocol Activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Limited Protocol Activities), Montvale, New Jersey
  - Memorial Sloan Kettering Cancer Center @ Suffolk-Commack (Consent only), Commack, New York
  - Memorial Sloan Kettering Westchester (Limited Protocol Activities), Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Nassau (Limited Protocol Activites), Rockville Centre, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org